CLINICAL TRIAL: NCT00470210
Title: Efficacy and Safety of High-dose Ribavirin (1600 mg/d) Boosted With Epoetin β (450 IU/kg/wk) in HIV/HCV Coinfected Patients Not Responding to Previous Treatment Regimens
Brief Title: Peginterferon Alfa-2a, Ribavirin and Epoetin β in Coinfected Patients HCV/HIV Not Responding to Previous Treatment Regimens
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Germans Trias i Pujol Hospital (Other)
Collaborators: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MORE; 2006-005554-74
Record Dates: First submitted 2007-05-04; First posted 2007-05-07 (Estimated); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: Hepatitis C; HIV Infections
Keywords: Ribavirin; non-responders; HCV co-infected patients; sustained virological response; Treatment Experienced
MeSH Terms: conditions — Hepatitis C; HIV Infections | interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Peginterferón alfa-2a (40 KD) (Pegasys®) 180 ug/week Ribavirin (Copegus®) 1600 mg/day Epoetin β (450 UI/kg/week)
  Interventions: Drug: Peginterferón alfa-2a (40 KD) (Pegasys®) 180 ug/week; Drug: Ribavirin (Copegus®) 1600 mg/day; Drug: Epoetin β (450 UI/kg/week)

INTERVENTIONS:
Drug: Peginterferón alfa-2a (40 KD) (Pegasys®) 180 ug/week — Peginterferón alfa-2a (40 KD) (Pegasys®) 180 ug/week
Drug: Ribavirin (Copegus®) 1600 mg/day — Ribavirin (Copegus®) 1600 mg/day
Drug: Epoetin β (450 UI/kg/week) — Epoetin β (450 UI/kg/week)

SUMMARY:
This trial will assess the sustained virologic response to treatment with peginterferon alfa-2a combined with high-dose ribavirin in human immunodeficiency virus (HIV)-infected patients with hepatitis C virus (HCV) genotype 1 or 4 coinfection and persistent transaminase elevations. These patients will have been nonresponders to previous regimens with peginterferon alfa and ribavirin therapy at a dosage of 800-1200 mg/d.

DETAILED DESCRIPTION:
The purpose in treating chronic HCV infection in HIV-coinfected individuals is to clear HCV-RNA antibodies and cure the infection. Studies have shown that high doses of ribavirin are associated with higher response rates than those achieved with ribavirin at dosages of 800-1200 mg/d.

The main aim of this trial is to assess the sustained virologic response to treatment with peginterferon alfa-2a plus high-dose ribavirin in HIV-infected patients coinfected with HCV genotypes 1 or 4 who have had persistent transaminase elevations and lack of response to previous treatment with peginterferon alfa and ribavirin at dosages of 800-1200 mg/d.

The second aim will be to measure changes in serum HCV-RNA titers and the percentage of patients achieving serum viral loads of < 50 IU/mL during treatment. Finally, we also intend to evaluate the safety of this treatment regimen.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected patients coinfected with HCV genotypes 1 or 4
* Persistent transaminase elevation
* Nonresponders to previous treatment with peginterferon alfa plus ribavirin at a dosage of 800-1200 mg/d.

Exclusion Criteria:

* Patients who abandoned treatment with peginterferon plus ribavirin before 12 weeks
* Patients with Child-Pugh B or C cirrhosis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-05; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Rate of sustained virologic response measured as serum HCV-RNA loads of < 50 IU/mL | 24 weeks after finishing treatment

SECONDARY OUTCOMES:
Changes in serum HCV-RNA titers | between baseline and 4, 8, 12, 24, and 48 weeks after start of treatment
Percentage of patients with serum HCV-RNA loads of < 50 IU/mL | at weeks 4, 8, 12, 24, and 48

CONTACTS AND LOCATIONS:
Overall Officials: Bonaventura Clotet, MD, PhD, Principal Investigator — Germans Trias i Pujol Hospital; Cristina Tural, MD, PhD, Principal Investigator — Germans Trias i Pujol Hospital
Locations (2):
- Spain (2):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital del Mar, Barcelona